CLINICAL TRIAL: NCT05559788
Title: A Study of Real-World Use of Selinexor, Daratumumab and Dexamethasone in Chinese Patients With Multiple Myeloma at First Relapse
Brief Title: Real-World Use of Selinexor, Daratumumab and Dexamethasone in Chinese Patients With Multiple Myeloma at First Relapse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fu chengcheng PhD (Other)
Responsible Party: Sponsor-Investigator, Fu chengcheng PhD, Principal Investigator, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Other Study IDs: SDd-MM06
Record Dates: First submitted 2022-08-11; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma at First Relapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Multiple Myeloma: Participants with MM who are first relapsed and will start treatment with selinexor, daratumumab and dexamethasone in a real-world clinical practice setting will be observed prospectively for approximately up to 1 year.

SUMMARY:
This is a single-arm, prospective, non-interventional, real-world study to observe and evaluate the efficacy and safety of selinexor in combination with daratumumab and dexamethasone in patients with multiple myeloma at first relapse.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, observational post-marketing surveillance study of selinexor, daratumumab and dexamethasone in participants with multiple myeloma (MM).

The study will assess the safety and effectiveness of selinexor in combination with daratumumab and dexamethasone (XDd) for first relapse MM patients under real-world conditions.

The study will enroll approximately 34 participants. The data will be prospectively collected, at our center from medical files and recorded into electronic case report forms (e-CRFs).

The overall duration of the study will be approximately 3 years. Data will be collected over and up to a 12 months-surveillance period (per participant) once enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. According to the multiple myeloma diagnostic criteria of the International Myeloma Working Group (IMWG), there is the initial diagnosis of multiple myeloma.
2. Subjects must have previously received 1 anti-myeloma regimens. Subjects must have documented disease progression
3. Age ≥18 years;
4. Life expectancy > 6 months;
5. patients should provide available clinical case files and/or detailed records of medical history, diagnosis and treatment information, and cooperate with clinical management;
6. Fertile women and men whose partner is of childbearing potential or pregnant should agree to practice complete abstinence or to use a condom during therapy and dose interruptions and for 90 days after the last treatment.

Exclusion Criteria:

1. Patients who are contraindicated as per product label of XDd;
2. Known positive for HIV or active hepatitis B or C or other infectious diseases;
3. Pregnancy or lactation;
4. Patients with a history of malignant tumor that may affect the implementation or results analysis of this study (except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, intramucosal carcinoma of the gastrointestinal tract in situ, and localized prostate cancer);
5. Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results;
6. Patients who are unsuitable for this study judged by clinicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with MM who who are first relapsed and will start treatment with selinexor, daratumumab and dexamethasone in a real-world clinical practice setting will be bserved prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 28 days after the last therapy
  ORR is defined as the percentage of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) based on the review of the myeloma response data assessed by International Myeloma Working Group (IMWG) criteria.